CLINICAL TRIAL: NCT02468700
Title: A Prospective, Multicenter, Randomized, Parallel-Arm, Bilateral, Double-Masked, Vehicle Controlled Feasibility Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Dry Eye
Brief Title: OTX-14-006: A Phase 2 Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-14-006
Record Dates: First submitted 2015-06-04; First posted 2015-06-11 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-DP (Experimental): OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use
  Interventions: Drug: Dexamethasone
- PV (Placebo Comparator): PV (placebo drug delivery vehicle)
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP
Other: Placebo Vehicle
  Arms: PV

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use when placed in the canaliculus of the eyelid for the treatment of the signs and symptoms of dry eye disease

ELIGIBILITY:
Inclusion Criteria:

* Had a known history of dry eye disease
* Had a minimal Corneal Fluorescein Staining Score and OSDI score in each eye

Exclusion Criteria:

* History of intraocular inflammation in either eye
* Use of the anti-inflammatory or immunomodulating agents ocular or systemic for the duration of the study
* Uncontrolled glaucoma or is on medications to treat glaucoma
* History of IOP spikes in either eye
* Active epiphora

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Vehicle: PV (placebo drug delivery vehicle)
Period: Overall Study
Arm/Group | OTX-DP | Placebo Vehicle
Started | 22 | 21
Completed | 20 | 19
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DP | Placebo Vehicle | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Full Range); unit: years] | 62.3 [41 to 84] | 62.5 [46 to 77] | 62.4 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Iris Color [Count of Participants; unit: Participants]
  Blue | 5 | 10 | 15
  Brown | 8 | 7 | 15
  Hazel | 7 | 3 | 10
  Green | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Corneal Fluorescein Staining
Description: National Eye Institute (NEI) Scale; Grade 0-3 for each region, 5 regions total (Total maximum score=15; 0=No staining)
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 22 | 21
units on a scale | 4.09 (2.671) | 5.05 (3.041)

2. Primary Outcome: Total Corneal Fluorescein Staining
Description: National Eye Institute (NEI) Scale; Grade 0-3 for each region, 5 regions total (Total maximum score=15; 0=No staining)
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 22 | 21
units on a scale | 4.64 (2.361) | 6.38 (3.278)

3. Primary Outcome: Total Conjunctival Lissamine Green Staining
Description: National Eye Institute (NEI) Scale; Grade 0-3 for each region, 6 regions total (Total maximum score=18; 0=No staining)
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 22 | 21
units on a scale | 4.36 (2.517) | 5.67 (4.199)

4. Primary Outcome: Total Conjunctival Lissamine Green Staining
Description: National Eye Institute (NEI) Scale; Grade 0-3 for each region, 6 regions total (Total maximum score=18; 0=No staining)
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 22 | 21
units on a scale | 6.41 (2.130) | 7.81 (3.642)

ADVERSE EVENTS:
Arm/Group | OTX-DP | Placebo Vehicle
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/21
Other Adverse Events (participants affected / at risk) | 15/22 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (N=22) | Placebo Vehicle (N=21)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (N=22) | Placebo Vehicle (N=21)
Adverse Events (General disorders) | 15 (24) | 11 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No